CLINICAL TRIAL: NCT01576588
Title: Study of Rituximab in Addition to Glucocorticoid in Pretreated Elderly or Unfit Patients With Chronic B Lymphocytic Leukemia
Brief Title: Rituximab in Pretreated Elderly or Unfit B-CLL Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. Med. Laimonas Griskevicius (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Med. Laimonas Griskevicius, Principal Investigator, Vilnius University
Organization: Vilnius University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LT-CLL-2s
Record Dates: First submitted 2012-03-09; First posted 2012-04-12 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia
Keywords: Chronic lymphocytic leukemia, relapsed, elderly or unfit patients, methylprednisolone, rituximab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Recurrence | interventions — Rituximab; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R-HDMP (Experimental): Rituximab (Rtx) antibody infusions will be administered on Day 1, 2, 3 (cycle 1) and Day 1 (cycles 2 to 4).
  Glucocorticoid (either Dexamethasone or Methyl-prednisolone) infusions will be administered on Days 1 to 3 (cycles 1-4(6)) and should precede the Rituximab infusion.
  Interventions: Drug: Rituximab; Drug: Glucocorticoid

INTERVENTIONS:
Drug: Rituximab — Rituximab (Rtx) antibody infusions will be administered on Day 1, 2, 3 (cycle 1) and Day 1 (cycles 2 to 4).
  Other Names: MabThera
Drug: Glucocorticoid — Glucocorticoid (either Dexamethasone or Methyl-prednisolone) infusions will be administered on Days 1 to 3 (cycles 1-4(6)) and should precede the Rituximab infusion.

SUMMARY:
The study will test the efficacy rituximab in addition to glucocorticoids for the treatment of B-CLL in elderly or unfit patients.

DETAILED DESCRIPTION:
Patient Population: Pretreated patients with symptomatic B-CLL 18-64 years of age with poor performance status or >/=65 years of age with any performance status.

Treatment: Up-to 4 cycles of glucocorticoid (Methylprednisolone or Dexamethasone) and Rituximab every 21 day.

Study Duration: The study period for each subject is expected to be 21 months. Subjects will receive up-to 4 cycles of IV infusion of Rituximab and Glucocorticoid. Maximum duration of treatment is expected to be 6 months. Subjects will complete scheduled visits not later than Study Month 21, thereafter they will enter into the long-term follow-up period. Subjects will be followed every 3 months for disease progression, initiation of subsequent leukemia treatment or survival.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of CD20 positive chronic B lymphocytic leukemia (BCLL) confirmed by biopsy or flow-cytometry.
* Previously treated patients with stage Rai I-IV and progressive disease (according to IWCLL 2008 guidelines).

Active B-CLL is defined by at least one of the following:

At least one of the disease related symptoms:

* Constitutional symptoms:
* Weight loss >10% within the previous 6 months;
* Fatigue (e.g., WHO performance status >/=2);
* Fever >/=38C >/=2 weeks without evidence of infection;
* Night sweats for more than 1 month without evidence of infection.
* Evidence of progressive marrow failure as manifested by development of, or worsening of, anemia and/or thrombocytopenia
* Autoimmune hemolysis and/or thrombocytopenia poorly responsive to corticosteroid therapy.
* Massive (i.e., >/=6 cm bellow left costal margin) or progressive or symptomatic splenomegaly.
* Massive lymphadenopathy or conglomerates (i.e., >/=10 cm in largest diameter) or progressive or symptomatic lymphadenopathy.
* Progressive lymphocytosis with an increase >50% over a 2-month period or an anticipated doubling time of less than 6 months. In patients with initial blood lymphocyte counts of less than 30x10^9/L LDT should not be used as a single parameter to define treatment indication. Marked hypogammaglobulinemia or the development of a monoclonal protein in the absence of any of the above criteria for active disease is not sufficient for protocol therapy.
* Either of the following:
* 18 years of age or older with impaired performance status (CIRS > 6) and /or
* 65 years of age or older with any performance status.
* Signed informed consent form.

Exclusion Criteria:

* Intolerance to exogenous protein or known severe reaction to the administration of Rituximab.
* Active infection.
* Cancer radiotherapy, biological therapy or chemotherapy within 3 weeks prior to Study Day 1.
* TBC or fungal infection within the past 6 months even if adequately controlled by treatment.
* Severe organ deficiency preventing the participation in the study.
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Study Day 1.
* Active peptic ulcer.
* Inadequately controlled diabetes mellitus.
* Suspected or confirmed B-CLL CNS disease.
* Known to be HIV positive.
* Difficult to control, uncooperative patients.
* Allergic disorders in need of chronic glucocorticoid therapy.
* Other oncological diseases requiring active treatment (except hormonal therapy).
* Pregnancy and breastfeeding.
* Patients of reproductive potential who are not using effective methods of contraception.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laimonas Griskevicius, MD, Principal Investigator — Hematology, Oncology and Transfusion Medicine Center, Vilnius University Hospital Santaros Klinikos
Locations (1):
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania

REFERENCES:
- [Background] Pileckyte R, Jurgutis M, Valceckiene V, Stoskus M, Gineikiene E, Sejoniene J, Degulys A, Zvirblis T, Griskevicius L. Dose-dense high-dose methylprednisolone and rituximab in the treatment of relapsed or refractory high-risk chronic lymphocytic leukemia. Leuk Lymphoma. 2011 Jun;52(6):1055-65. doi: 10.3109/10428194.2011.562572. PMID 21599591
- [Background] Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating MJ, Montserrat E, Rai KR, Kipps TJ; International Workshop on Chronic Lymphocytic Leukemia. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 guidelines. Blood. 2008 Jun 15;111(12):5446-56. doi: 10.1182/blood-2007-06-093906. Epub 2008 Jan 23. PMID 18216293
- [Result] Pileckyte R, Valceckiene V, Stoskus M, Matuzeviciene R, Sejoniene J, Zvirblis T, Griskevicius L. Dose Intensive Rituximab and High-Dose Methylprednisolone in Elderly or Unfit Patients with Relapsed Chronic Lymphocytic Leukemia. Medicina (Kaunas). 2019 Oct 29;55(11):719. doi: 10.3390/medicina55110719. PMID 31671877

RESULTS

PARTICIPANT FLOW:
Groups:
- R-HDMP: Rituximab (Rtx) antibody infusions will be administered on Day 1, 2, 3 (cycle 1) and Day 1 (cycles 2 to 4).
  Glucocorticoid (either Dexamethasone or Methyl-prednisolone) infusions will be administered on Days 1 to 3 (cycles 1-4(6)) and should precede the Rituximab infusion.
  Rituximab: Rituximab (Rtx) antibody infusions will be administered on Day 1, 2, 3 (cycle 1) and Day 1 (cycles 2 to 4).
  Glucocorticoid: Glucocorticoid (either Dexamethasone or Methyl-prednisolone) infusions will be administered on Days 1 to 3 (cycles 1-4(6)) and should precede the Rituximab infusion.
Period: Overall Study
Arm/Group | R-HDMP
Started | 25
Completed | 23
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | R-HDMP
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 25
Age, Continuous [Median (Full Range); unit: years] | 73 [65 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Lithuania | 25

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Overall response rate (ORR) is defined according to International Workshop on Chronic Lymphocytic Leukemia (iwCLL 2008) guidelines, as the proportion of patients achieving complete response (CR), CR with minimal residual disease (MRD) negativity (complete molecular remission), nodular partial remission (nPR) and partial response (PR).
Time Frame: 3 months +/- 2 weeks after the last treatment cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | R-HDMP
Number analyzed (Participants) | 25
Participants | 7

2. Secondary Outcome: Progression Free Survival
Description: Progression free survival (PFS) will be defined as the interval from entry into the study to disease progression or death.
Time Frame: up to 12 months
Measure: Median (Full Range); unit: months
Arm/Group | R-HDMP
Number analyzed (Participants) | 25
months | 11 [10 to 12]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events NCI CTCAE, version 4.0. Hematological toxicity was evaluated according to IWCLL 2008 guidelines.
Time Frame: 6 months.
Population: Patient, who experienced any AE - 23.
Measure: Count of Participants; unit: Participants
Arm/Group | R-HDMP
Number analyzed (Participants) | 25
Participants | 23

4. Secondary Outcome: Overall Survival
Description: Overall survival (OS) will be defined as the interval from date of randomization until the date of death from any cause, assessed up to 100 months.
Time Frame: from date of randomization until the date of death from any cause, assessed up to 100 months
Measure: Median (Full Range); unit: months
Groups:
- R-HDMP: Rituximab (Rtx) antibody infusions will be administered on Day 1, 2, 3 (cycle 1)...
Arm/Group | R-HDMP
Number analyzed (Participants) | 25
months | 68 [47 to 89]

ADVERSE EVENTS:
Arm/Group | R-HDMP
Serious Adverse Events (participants affected / at risk) | 9/25
Other Adverse Events (participants affected / at risk) | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-HDMP (N=25)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) — Febrile neutropenia
Extrasystolia (Cardiac disorders) | 1 (1)
Orfarin overdosage (Social circumstances) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Diarea (Gastrointestinal disorders) | 2 (2)
Upper pulmonary infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Left femur cervical stress fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Renal insufficiency (Renal and urinary disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | R-HDMP (N=25)
Hyperglycemia (Endocrine disorders) | 2 (3)
Hypertention (Cardiac disorders) | 4 (13)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chest discomfort/pain (Cardiac disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (2)
Fever (Infections and infestations) | 3 (5)
Hypokalemia (Metabolism and nutrition disorders) | 15 (26)
hypomagnesemia (Metabolism and nutrition disorders) | 2 (3)
Insomnia (Nervous system disorders) | 3 (3)
Leg edema (Blood and lymphatic system disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No